CLINICAL TRIAL: NCT03351530
Title: Development of a Molecular Diagnosing Platform for Monitoring Oral Hygiene in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: General Biologicals Corporation (Industry)
Collaborators: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 16CT044be
Record Dates: First submitted 2017-11-09; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus; Periodontal Diseases
MeSH Terms: conditions — Diabetes Mellitus; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Pre-diabetes
- Diabetes
- Diabetes with periodontal disease
- Periodontal patient
- Healthy person

SUMMARY:
More than ninety percent of adults in Taiwan are suspected to carry periodontal disease, which causes bad breath, swollen and bleeding gums, plaque and even tooth loss. Half of the patients, however, are ignorance these clinical syndromes because of no obvious pain. A lot of researches show that periodontal disease is related to diabetes mellitus. Periodontal disease causes rise of blood sugar, and more than 3 times as diabetes mellitus patients as healthy people have serious periodontal disease.In this study, the investigators collect periodontal pocket and saliva samples of participants, and selecting six periodontal disease-associated bacteria strains, including Porphyromonas gingivalis (Pg), Fusobacterium nucleatum (Fn), Actinobacillus actinomycetemcomitans (Aa), Treponema denticola (Td), Prevotella intermedia (Pi) and Tannerella forsythia (Tf) as diagnostic markers. Participants will get bacteriostasis mouthwash at mouth 2. The investigators will compare the differences of blood biochemistry value and oral bacteria strains after using the mouthwash.Using real-time PCR and MALDI Biotyper, the investigators will establish the database of oral microorganisms in diabetes mellitus patients, providing periodontal disease clinical markers of high-risk groups and the basis for personal medicine of therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion condition of diabetes:

1. HbAlC≧6.5%
2. Glucose(AC)≧126 mg/dL
3. 2-h PG≧200mg/dL during an OGTT
4. In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose≧200mg/dL 2. Inclusion condition of periodontal disease

(1) 16 natural teeths and 6 front teeth at lesat (2) Periodontal pocket≧7 mm, and radiographic bone loss≧30%

Exclusion Criteria:

1. People who have oral lesion, dental braces, denture, mouthwash allergy, or serious systemic disease
2. People who have ever eaten antibiotics and Anti-inflammatory drugs over the last 6 months
3. People who have ever eaten Immunosuppressive drugs, antiepileptic drugs, antihypertensive drugs, or anticoagulant
4. Pregnant women or the woman who eat birth control pills

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Diabetes:
  1. HbAlC≧6.5%
  2. Glucose(AC)≧126 mg/dL
  3. 2-h PG≧200mg/dL during an OGTT
  4. In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose≧200mg/dL 2. Periodontal disease
  (1) 16 natural teeths and 6 front teeth at lesat (2) Periodontal pocket≧7 mm, and radiographic bone loss≧30%
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-12-09 (Estimated); Study Completion 2019-02-09 (Estimated)

PRIMARY OUTCOMES:
The change of glucose (AC) between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of glucose (AC) in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash.
The change of HbAlC between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of HbAlC in % with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash.
The change of cholesterol total between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of cholesterol total in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of triglyceride between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of triglyceride in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of LDL between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of LDL in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of HDL between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of HDL in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of uric acid between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of uric acid in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of GPT between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of GPT in U/L with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of creatinine between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of creatinine in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of micro-albumin between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of micro-albumin in mg/L with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash
The change of hs-CRP between diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 6 month
  To compare the value of hs-CRP in mg/dL with diabetes mellitus patients, periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash

CONTACTS AND LOCATIONS:
Locations (1):
- General Biologicals Corporation, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagaoka K, Yanagihara K, Morinaga Y, Nakamura S, Harada T, Hasegawa H, Izumikawa K, Ishimatsu Y, Kakeya H, Nishimura M, Kohno S. Prevotella intermedia induces severe bacteremic pneumococcal pneumonia in mice with upregulated platelet-activating factor receptor expression. Infect Immun. 2014 Feb;82(2):587-93. doi: 10.1128/IAI.00943-13. Epub 2013 Nov 18. PMID 24478074
- [Background] Suzuki J, Imai Y, Aoki M, Fujita D, Aoyama N, Tada Y, Wakayama K, Akazawa H, Izumi Y, Isobe M, Komuro I, Nagai R, Hirata Y. Periodontitis in cardiovascular disease patients with or without Marfan syndrome--a possible role of Prevotella intermedia. PLoS One. 2014 Apr 18;9(4):e95521. doi: 10.1371/journal.pone.0095521. eCollection 2014. PMID 24748407
- [Background] Hajishengallis G. Periodontitis: from microbial immune subversion to systemic inflammation. Nat Rev Immunol. 2015 Jan;15(1):30-44. doi: 10.1038/nri3785. PMID 25534621
- [Background] Grossi SG, Genco RJ. Periodontal disease and diabetes mellitus: a two-way relationship. Ann Periodontol. 1998 Jul;3(1):51-61. doi: 10.1902/annals.1998.3.1.51. PMID 9722690
- [Background] Lalla E, Papapanou PN. Diabetes mellitus and periodontitis: a tale of two common interrelated diseases. Nat Rev Endocrinol. 2011 Jun 28;7(12):738-48. doi: 10.1038/nrendo.2011.106. PMID 21709707